CLINICAL TRIAL: NCT03549598
Title: d68Ga-DOTATATE PET/CT Assessment of Cardiac Sarcoidosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John P. Bois, M.D., Assistant Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-000393
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Cardiac Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTATATE PET/CT (Experimental): 68Ga-DOTATATE PET/CT scan, 18FDG PET/CT scan and 13NH3 PET/CT scan will be performed on each subject
  Interventions: Drug: 68Ga-DOTATATE PET/CT; Drug: 18FDG PET/CT scan; Drug: 13NH3 PET/CT scan

INTERVENTIONS:
Drug: 68Ga-DOTATATE PET/CT — 5.4 mCi of 68Ga-DOTATATE will be administered by intravenous route.
Drug: 18FDG PET/CT scan — This scan will be performed as part of the planned clinical care for the patient. Dose of 18FDG will be administered intravenously in accordance with the institutional policy and accepted norms. CT attenuation scan will also be performed as part of this examination per institutional protocol.
Drug: 13NH3 PET/CT scan — This scan will be performed as part of the planned clinical care for the patient. Dose of 13NH3 will be administered intravenously in accordance with the institutional policy and accepted norms. CT attenuation scan will also be performed as part of this examination per institutional protocol.

SUMMARY:
The Researchers are trying to determine if 68Ga-DOTATATE PET/CT imaging will have a similar accuracy as 18FDG PET/CT in diagnosing cardiac sarcoidosis and if it will be able to do so without the need for complex patient dietary preparation that is required with 18FDG PET/CT.

DETAILED DESCRIPTION:
Prospective study of 15 consecutive patients with suspected or newly diagnosed cardiac sarcoidosis (CS) who are referred for a clinically indicated 18FDG (and 13NH3) PET/CT scan for cardiac sarcoidosis (CS) will be approached to undergo a 68Ga-DOTATATE PET/CT scan. Comparison will then be made between the 68Ga-DOTATATE PET/CT and the 18FDG and 13NH3 PET/CT to determine if 68Ga-DOTATATE detects CS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Referred for clinically indicated 18FDG PET/CT scan for cardiac sarcoidosis (CS)

Exclusion Criteria:

* Pregnant
* Unable or unwilling to give consent for 68Ga-DOTATATE PET/CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Bois, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- 68Ga-DOTATATE PET/CT: 68Ga-DOTATATE PET/CT scan, 18FDG PET/CT scan and 13NH3 PET/CT scan were be performed on each subject
  68Ga-DOTATATE PET/CT: 5.4 mCi of 68Ga-DOTATATE were administered by intravenous route.
  18FDG PET/CT scan: This scan was performed as part of the planned clinical care for each subject. Dose of 18FDG was administered intravenously in accordance with the institutional policy and accepted norms. CT attenuation scan was also performed as part of the examination per institutional protocol.
  13NH3 PET/CT scan: This scan was performed as part of the planned clinical care for each subject. Dose of 13NH3 was administered intravenously in accordance with the institutional policy and accepted norms. CT attenuation scan was also be performed as part of this examination per institutional protocol.
Period: Overall Study
Arm/Group | 68Ga-DOTATATE PET/CT
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 68Ga-DOTATATE PET/CT
Number analyzed (Participants) | 15
Age, Continuous [Median (Standard Deviation); unit: years] | 70 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: 68Ga-DOTATATE Uptake With Cardia Sarcoidosis (CS)
Description: The number of subjects with areas of abnormal myocardial increased focal uptake
Time Frame: 3 days
Population: Unreliable or uninterpretable data due to background uptake on 68Ga-DOTATATE scans. Data not obtained and was not analyzed
Arm/Group | 68Ga-DOTATATE PET/CT
Number analyzed (Participants) | 0

2. Primary Outcome: 18FDG Uptake With Cardia Sarcoidosis (CS)
Description: The number of subjects with areas of abnormal myocardial increased focal uptake on 18FDG scan
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | 68Ga-DOTATATE PET/CT
Number analyzed (Participants) | 15
Participants | 9

3. Primary Outcome: 13NH3 PET/CT Uptake With Cardia Sarcoidosis (CS)
Description: The number of subjects with areas of perfusion deficits on 13NH3 PET/CT scan
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | 68Ga-DOTATATE PET/CT
Number analyzed (Participants) | 15
Participants | 8

4. Secondary Outcome: Physician Confidence in Study Interpretation
Description: A Physician survey will be conducted for those cardiac imagers assessing both the DOTATATE and FDG studies to determine their confidence level in interpreting the studies and if one study was easier to interpret than the other
Time Frame: 2 days
Population: Unreliable or uninterpretable data due to background uptake on 68Ga-DOTATATE scans. Data unable to obtain and was not analyzed
Arm/Group | 68Ga-DOTATATE PET/CT
Number analyzed (Participants) | 0

5. Secondary Outcome: Subject Satisfaction
Description: A patient survey will be conducted after each subject has undergone both the DOTATE and the FDG scans. Patient satisfaction will be measured by the question, "Which study did you prefer?" Subject to circle one of the following: 18FDG, 68Ga-DOTATATE or Equal
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | 68Ga-DOTATATE PET/CT
Number analyzed (Participants) | 15
Participants
  18FDG | 0
  68GA-DOTATATE | 13
  Equal | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to through end of study (completion of last scan), approximately 3 days
Groups:
- 68Ga-DOTATATE PET/CT: 68Ga-DOTATATE PET/CT scan, 18FDG PET/CT scan and 13NH3 PET/CT scan were be performed on each subject
  68Ga-DOTATATE PET/CT: 5.4 mCi of 68Ga-DOTATATE were administered by intravenous route.
- 18FDG PET/CT: 68Ga-DOTATATE PET/CT scan, 18FDG PET/CT scan and 13NH3 PET/CT scan were be performed on each subject
  18FDG PET/CT scan: This scan was performed as part of the planned clinical care for each subject. Dose of 18FDG was administered intravenously in accordance with the institutional policy and accepted norms. CT attenuation scan was also performed as part of the examination per institutional protocol.
- 13NH3 PET/CT": 68Ga-DOTATATE PET/CT scan, 18FDG PET/CT scan and 13NH3 PET/CT scan were be performed on each subject
  13NH3 PET/CT scan: This scan was performed as part of the planned clinical care for each subject. Dose of 13NH3 was administered intravenously in accordance with the institutional policy and accepted norms. CT attenuation scan was also be performed as part of this examination per institutional protocol.
Arm/Group | 68Ga-DOTATATE PET/CT | 18FDG PET/CT | 13NH3 PET/CT"
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 68Ga-DOTATATE PET/CT (N=15) | 18FDG PET/CT (N=15) | 13NH3 PET/CT" (N=15)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Unreliable or uninterpretable data due to background uptake on 68Ga-DOTATATE scans

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT03549598/Prot_SAP_000.pdf